CLINICAL TRIAL: NCT05685095
Title: Impact de Programmes de Marche Active Sur la Marche en Situation de Vie Quotidienne et la qualité de Vie Dans la Maladie de Parkinson
Brief Title: Programmes de Marche Active et qualité de Vie Dans la Maladie de Parkinson
Acronym: ACTI-PARK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: personnel involved in clinical trial will not be available to conduct the research
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 38RC22.0105_ACTI-PARK; 2022-A00678-35 (Other: ID RCB)
Record Dates: First submitted 2022-09-01; First posted 2023-01-13 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: adapted physical activity; gait; quality of life; actimetry; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers involved in data collection and in data analysis will be blinded with regard to the patients' group allocation. Randomization will be performed by an operator not otherwise involved in the study, under the RED-Cap application.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill walking (Experimental): The training program will last 12 weeks and consist of treadmill walking. The duration of the walking bouts (and pauses), and the speed of the belt will be adjusted as needed following the patients' progress. Music will be added as suited to boost motivation and support regular cadence. All training sessions will be supervised.
  Interventions: Behavioral: Physical training
- Nordic walking (Experimental): The training program will last 12 weeks and consist of Nordic walking, taught and supervised by an adapted physical activity teacher. The session will be carried out outside, weather permitting. When possible, training will gather 2 to 4 patients for group emulation. The duration of the walking bouts (and pauses) will be adjusted to follow the patients' progress.
  Interventions: Behavioral: Physical training

INTERVENTIONS:
Behavioral: Physical training — Supervised gait training program 3 times a week, 12 weeks

SUMMARY:
The aim of this randomized controlled pilot trial is to assess the impact of different gait rehabilitation programs on the level of physical activity and gait in daily life in patients with Parkinson's disease (PD).

Two groups of 25 patients with PD will benefit from one of two gait training programs (treadmill vs. nordic walking), 3 times a week for 12 weeks. Activity level and number of steps will be remotely recorded over 7 days before, at the end, 3 and 6 months after the end of the program. Quality of life will be recorded at each time point.

The impact of the gait programs on the patients' level of daily activity will be examined, comparing the changes brought about by the two programs, taking into account the modulating influence of age and cognitive function.

Gait under conditions of daily life will be compared to gait parameters collected in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, diagnosed for at least 2 years,
* Medical treatment (if any) unchanged in the past 4 weeks at least
* Hoehn & Yahr score < 3
* Montreal cognitive assessment (MOCA) score between 20 and 30
* Able to understand the aim and methods of the study and provide signed informed consent-

Exclusion Criteria:

* Atypical parkinsonian syndrome
* Cardiovascular pathology preventing moderate physical exercise
* Orthostatic hypotension
* Any condition (other than PD) interfering with gait
* pregnant or nursing

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Changes in daily energy expenditure | recording 7 days in a row, at 3 months, 6 months and 9 months.
  Evolution over time of the daily energy expenditure together with number of steps, as recorded using an actimeter worn at the belt.

SECONDARY OUTCOMES:
Evolution of gait parameters | 3 months, 6 months and 9 months.
  Evolution over time of spatio-temporal gait parameters recorded during a gait test in the laboratory.
Evolution of exercise functional capacity | 3 months, 6 months and 9 months.
  Evolution over time of the patients' performance at the 6 minutes walk test
Evolution over time of the Parkinson's Disease Questionnaire-39 scale score. | 3 months, 6 months and 9 months.
  Evolution of quality of life as measured using the PDQ.39 scale. Summed item scores expressed as percent. Min 0 Max 100.
Evolution over time of the Parkinsons' Disease Fatigue Scale score. | 3 months, 6 months and 9 months.
  Evolution of fatigue as measured using the PD Fatigue scale. Min 0. Max 80. Greater score means greater fatigue
Adherence to the training program | 3 months
  number of training sessions attended

CONTACTS AND LOCATIONS:
Overall Officials: Moro Elena, MD PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No